CLINICAL TRIAL: NCT04162145
Title: BRIDGE Device for Symptoms of Opioid Withdrawal: A Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: BRIDGE Device for Treatment of Opioid Withdrawal
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 pandemic
Sponsor: BrightView LLC (Industry)
Collaborators: Innovative Health Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7454-JACraven
Record Dates: First submitted 2019-11-07; First posted 2019-11-14 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Opioid Withdrawal; Pain; Craving
Keywords: opioid withdrawal; opioid; pain; craving; NSS-2 BRIDGE; percutaneous electrical nerve field stimulator (PENFS)
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Two groups will be studied: one group using active BRIDGE devices and one using sham or inactive devices.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be randomly assigned to one of the 2 treatment groups in equal ratio. Randomization will be done centrally using a randomized block design, with blocks of 4 using the Pqantadosi Randomization software. There will be a randomization table provided to the person dispensing the devices. The unblinded, lead research coordinator will keep the data in a secure database and will not be involved in any of the patient recruitment or study procedures. All other research coordinators, investigators, and nurses involved will be blinded to group allocation. In general, the study biostatisticians and the person dispensing will be the only people un-blinded throughout the duration of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active Device (Active Comparator): Patients in the Active Device arm will receive placement of an active BRIDGE device.
  Interventions: Device: Active BRIDGE device placement
- Sham Device (Sham Comparator): Patients in the Sham Device arm will receive placement of an inactive, or sham, BRIDGE device. The inactive device will be identical in appearance to the active device but will have no electrical current.
  Interventions: Device: Inactive BRIDGE device placement

INTERVENTIONS:
Device: Active BRIDGE device placement — The active BRIDGE device will be placed by a blinded medical provider. The severity of opioid withdrawal signs and symptoms will be assessed with the COWS, pain and cognitive functioning tests at several time points. Patients will be dosed with buprenorphine at the blinded provider's discretion. Supportive medications to help manage signs and symptoms of opioid withdrawal will NOT be allowed for one hour after the first dose of buprenorphine. Subjects will be asked to return to clinic for additional visits based on the clinic standard of care. Subjects will be reassessed using COWS, OCS and VAS at each subsequent visit, or remotely (via phone) when unrequired to return to clinic during the 5-day trial. The device will be removed at the clinic visit on Day 5 and disposed of in a sharps container. If the patient cannot come back on day 5, they will be instructed to remove the device at home and bring it back at the next clinic appointment for proper disposal.
  Arms: Active Device
Device: Inactive BRIDGE device placement — The inactive or sham BRIDGE device will be placed by a blinded medical provider. The severity of opioid withdrawal signs and symptoms will be assessed with the COWS, pain and cognitive functioning tests at several time points. Patients will be dosed with buprenorphine at the blinded provider's discretion. Supportive medications to help manage signs and symptoms of opioid withdrawal will NOT be allowed for one hour after the first dose of buprenorphine. Subjects will be asked to return to clinic for additional visits based on the clinic standard of care. Subjects will be reassessed using COWS, OCS and VAS at each subsequent visit, or remotely (via phone) when unrequired to return to clinic during the 5-day trial. The device will be removed at the clinic visit on Day 5 and disposed of in a sharps container. If the patient cannot come back on day 5, they will be instructed to remove the device at home and bring it back at the next clinic appointment for proper disposal.
  Arms: Sham Device

SUMMARY:
The purpose of this study is to prospectively evaluate the effectiveness of the NSS-2 BRIDGE device in reducing the signs and symptoms of acute opioid withdrawal when compared to placebo.

DETAILED DESCRIPTION:
The BRIDGE device is a novel, non-pharmacological, non-invasive, auricular percutaneous electrical nerve field stimulator (PENFS) that is thought to significantly reduce pain and modulate the autonomic nervous system through application to branches of Cranial Nerves V, VII, IX, and X, as well as branches of the occipital nerves identified by transillumination. The novelty of this device is in the use of alternating current and higher voltage stimulation over a large field in the external ear that allows access into central brain regions involved in fear and pain modulation. This device has been approved by the United States Food and Drug Administration (FDA) to treat the symptoms of opioid withdrawal.

In this study, the BRIDGE device will be compared to a "sham" (inactive) device. The sham device will be identical in appearance to the active device but will have no electrical current. Neither the patient or the study doctor/study staff will know whether an active or inactive device is being used during the study (double-blind).

The effectiveness of the device in reducing signs and symptoms of opioid withdrawal will be measured by:

* Assessing the severity of opioid withdrawal symptoms pre and post device placement for a period of 5 days.
* Assessing improvements in pain, craving and cognition pre and post device placement for a period of 5 days.

The investigators hypothesize that treatment with the BRIDGE device will have a significant and profound effect on decreasing opioid withdrawal scores compared to sham. The investigators also hypothesize that the BRIDGE device will have a significant and profound effect on decreasing pain and craving scores quickly in the two hours following application as well as the ensuing 4-5 days, and will demonstrate improvement in memory and executive function compared to sham treatment.

Patients going through acute opioid withdrawal will be assessed for the severity of opioid withdrawal using the Clinical Opioid Withdrawal Scale (COWS). Additional demographic data will be collected at presentation including age, sex, duration of opioid misuse, types of medications or illicit drugs used as well as the presence of other medical conditions. After the severity of opioid withdrawal is established (COWS score ≥10), subjects will be randomized in blinded fashion. Once the patient is consented, a visual analog scale (VAS) for pain and an opioid craving scale (OCS) will be completed. Baseline cognitive function will be measured with the Stroop test using the CNS Vital Signs (CNSVS) in-office neurocognitive testing software (https://www.cnsvs.com/index.html). This instrument measures executive function. The test takes approximately 4 minutes to administer and will be performed at the same intervals as COWS score, pain and craving assessments before and after device placement.

The severity of opioid withdrawal signs and symptoms will be assessed with the COWS at several time points: 1) pre-device placement, 2) 1-hour post placement of sham or active device, 3) two hours post placement (approximately one hour after first dose of buprenorphine), 4) at subsequent follow-up in clinic on day 2 and 5) at final follow-up in clinic on day 5 prior to removal of device. The visual analogue pain and craving scale will also be administered at intervals to monitor patient comfort: 1) pre-device placement, 2) 1-hour post placement of sham or active device, 3) two hours post placement (approximately one hour after first dose of buprenorphine),4) at subsequent follow-up in clinic on day 2, 5) in clinic or remotely (via phone) on days 3 and 4, and 6) at final follow-up in clinic on day 5 prior to removal of device. Assessment of cognitive function (CNSVS) will be recorded at 1) pre-device placement, 2) 1-hour post placement of sham or active device, and 5) at final follow-up in clinic on day 5 prior to removal of device.

One hour following placement of either sham or active device, the patients will be given the first dose of buprenorphine with a starting dose of 2, 4 or 8 mg at the blinded provider's discretion based on BMI, patient previous experience with BUP, patient apprehension or other factors. Adjustments to this dose will not be made for at least an hour after receiving the first dose but the providing clinician may order additional buprenorphine after one hour as indicated by initial response, previous experience, presence of precipitated clinical opioid withdrawal scale (COWS) and BMI. Subsequent adjustments will be made based on the blinded provider's discretion and patient needs and comfort as per clinic standard. Ancillary (supportive) medications to help manage signs and symptoms of opioid withdrawal will NOT be allowed for one hour after the first dose of buprenorphine. Following the first hour, symptom control medications including ibuprofen, clonidine, ondansetron, loperamide, and acetaminophen may be furnished or prescribed. A medication log will be provided to track usage of this modality. Subjects will remain blinded and keep the device on for 5 days regardless of randomization status. Subjects will be asked to return to clinic for additional induction visits based on the clinic standard of care which will be Day 2 and in some cases Days 3 & 4. In order to monitor whether neurostimulation with the BRIDGE has any added benefit for patients on outpatient opioid agonist therapy, subjects (regardless of active or placebo) will be reassessed using OCS and VAS at each subsequent visit, or remotely (via phone) when unrequired to return to clinic, during the 5-day trial.

Overall, the study will have very little deviation from the current standard of practice to treat substance use disorder (SUD), with the exception of the first hour of medical management which will be effected without buprenorphine or symptom control medications, and the second hour during which symptom control medications will not be used. Current standard of practice in the clinical setting is to give the first dose of buprenorphine on Day 1 after initial screening, followed by a second or third dose prior to discharge home. Patients will be sent home and monitored as outpatients and asked to return to clinic within 2-5 days. The current study will not deviate from clinical practice after Day 1 with the exception of having either the BRIDGE device or sham device for 5 days. The device will be removed at the clinic visit on Day 5 and disposed of in a sharps container. If the patient cannot come back on day 5, they will be instructed to remove the device at home and bring it back at the next clinic appointment for proper disposal. If at any time the patient wishes to discontinue the BRIDGE device and receive standard treatment for opioid withdrawal outside the study, he/she will be allowed to do so.

All data collected will be entered into a Redcap database for analysis. All collected data will be de-identified and samples will only have a unique identifier that will link the unique identifier with the patient's name. Results of the COWS and pain VAS scores, OCS and CNSVS assessments at the respective time points will be tabulated and analyzed. Upon completion of each patient's treatment with the device (sham or active), patients will be asked if they thought they had an active or inactive device.

Participants will also be asked to respond to the following:

• Does [the participant] want an active, functioning device to be placed prior to going home today? (yes/no)

And the following questions will be scored by the participants on a 7 point Likert scale:

1. How useful does [the participant] think the BRIDGE Device was for [the participant] overall in [the participant's] treatment?
2. What is [the participant]'s impression of the effectiveness of the BRIDGE Device to treat [the participant's] symptoms of withdrawal?
3. How satisfied is [the participant] with how the BRIDGE device worked for [the participant]?
4. How likely is [the participant] to use the device again if [the participant] has symptoms of withdrawal?

Results will be tabulated and analyzed descriptively. Analysis will also include differences in dosing of buprenorphine as well as usage of other symptom control medications and continued engagement in recovery treatment at 5- and 30-days post-device placement. If the patient does not return to the clinic at the 5- and 30-day scheduled appointment as dictated by clinic standard practice, a phone call will be made to assess whether the patient is still engaged in a recovery program.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be 18 years or older who speak English and meet criteria for opioid use disorder based on the Diagnostic and Statistical Manual of Mental Disorders-5.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-06-23 (Actual); Study Completion 2020-06-23 (Actual)

PRIMARY OUTCOMES:
Comparison of change from baseline of Clinical Opiate Withdrawal Scale (COWS) scores between active BRIDGE device group and sham BRIDGE device group at one hour | 3 months
  The primary outcome is comparison of change from baseline of the Clinical Opiate Withdrawal Scale (COWS) scores( score: 5-12=Mild; 13-24=Moderate; 25-36=Moderately Severe; More than 36=Severe Withdrawal) between active BRIDGE device group and sham BRIDGE device group at one hour. The two groups will be compared using a two-sided two sample t-test at an alpha of 0.001 at an interim analysis of the first 24 completing and at an alpha of 0.049 after 50 have completed.
  For all the efficacy parameters (e.g. Clinical Opiate Withdrawal Scale, Visual Analog Scale, Opioid Craving Scale and the Stroop test using CNS Vital Signs) the descriptive statistics will include N, mean median, standard error (SE), minimum and maximum or percentage and exact Clopper Pearson 95% confidence interval.

SECONDARY OUTCOMES:
Comparison of change from baseline of Clinical Opiate Withdrawal Scale (COWS) scores between active BRIDGE device group and sham BRIDGE device group over time for up to 3 months | 3 months
  As a secondary analysis the investigators will examine the change over time of the Clinical Opiate Withdrawal Scale (COWS) scores between groups using a mixed-effects model repeated measures (MMRM) analysis incorporating treatment period data up to 3 months.
  The effects in the model will include the baseline score, treatment groups, visit, treatment-by-visit interaction and baseline-by-visit interaction. Visit week will be treated as the repeated variable within a patient. Patient, treatment, and visit will be treated as class variables. Unstructured covariance matrix will be used initially, and additional types (e.g., auto- regression, Toeplitz, CS, etc.) will be tried to assess the robustness of the unstructured matrix. Comparison between treatments will be based on contrasts of least square treatment means at each week of interest. Least square means, standard errors, and 95% confidence intervals (CI) of treatment difference will be reported for the two groups.
Comparison of change from baseline of pain Visual Analog Scale (VAS) scores between active BRIDGE device group and sham BRIDGE device group over time for up to 3 months | 3 months
  As a secondary analysis the investigators will examine the change over time of the pain Visual Analog Scale (VAS) scores (0= not at ll, 10=extremely) between groups using a mixed-effects model repeated measures (MMRM) analysis incorporating treatment period data up to 3 months.
Comparison of change from baseline of Opioid Craving Scale (OCS) scores between active BRIDGE device group and sham BRIDGE device group over time for up to 3 months | 3 months
  As a secondary analysis the investigators will examine the change over time of the Opioid Craving Scale (OCS) scores (0= not at all, 10=extremely) between groups using a mixed-effects model repeated measures (MMRM) analysis incorporating treatment period data up to 3 months.
  The effects in the model will include the baseline score, treatment groups, visit, treatment-by-visit interaction and baseline-by-visit interaction. Visit week will be treated as the repeated variable within a patient. Patient, treatment, and visit will be treated as class variables. Unstructured covariance matrix will be used initially, and additional types (e.g., auto- regression, Toeplitz, CS, etc.) will be tried to assess the robustness of the unstructured matrix. Comparison between treatments will be based on contrasts of least square treatment means at each week of interest. Least square means, standard errors, and 95% confidence intervals (CI) of treatment difference will be reported for the two groups.
Comparison of change from baseline of cognition Stroop test scores using CNS Vital Signs software between active BRIDGE device group and sham BRIDGE device group over time for up to 3 months | 3 months
  As a secondary analysis the investigators will examine the change over time of cognitive function measured by the Stroop test (CNS Vital Signs) between groups using a mixed-effects model repeated measures (MMRM) analysis incorporating treatment period data up to 3 months. The test has three parts. In the first, the words RED, YELLOW, BLUE and GREEN (printed in black) appear at random on the screen, and the subject presses the space bar as soon as he or she sees the word. This generates a simple reaction time score.The subject is asked to press the space bar when the color of the word matches what the word says. This generates a complex reaction time score. In the third part, the subject is asked to press the space bar when the color of the word does not match what the word says. This part also generates a complex reaction time score, called the "Stroop reaction time.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Brightview LLC, Cincinnati, Ohio
  - BrightView, Cincinnati, Ohio

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/45/NCT04162145/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/45/NCT04162145/ICF_001.pdf